CLINICAL TRIAL: NCT01296698
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 26-Week Trial to Measure the Efficacy and Safety of a Novel Nicotine Replacement Therapy in Smokers in a Naturalistic Environment
Brief Title: Study to Determine if a New Nicotine Replacement Therapy Can Safely Help Smokers to Quit Smoking
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to a technical issue (randomization error).
Sponsor: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry)
Collaborators: McNeil AB (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A6431112
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0 mg Oral NRT, up to 4 times per hour for 12 weeks
  Interventions: Drug: Placebo
- Nicotine (Experimental): 1 mg Oral NRT, up to 4 times per hour for 12 weeks
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Placebo — Dosage Form: Oral NRT; Dose: 0 mg; Frequency: up to 4 times per hour; Duration: 12 weeks
  Other Names: Not marketed
  Arms: Placebo
Drug: Nicotine — Dosage Form: Oral NRT; Dose: 1 mg;Frequency: up to four times per hour; Duration:12 weeks
  Other Names: Not yet marketed
  Arms: Nicotine

SUMMARY:
This study is to see if a new nicotine replacement therapy safely helps people to quit smoking if it is used the way it would be if it were sold at the pharmacy and used at home. Approximately 1500 subjects will be enrolled into the study. The study will require participants to use the treatment for 12 weeks and there will be a 14-week follow-up period. The study will be conducted in approximately 20 pharmacies across the United States.

At the first visit to the pharmacy, participants will be asked some questions to see if they are eligible to participate. Participants will be asked to sign a consent form if they agree to participate. Participants will answer some more questions, and blow into a machine to measure their carbon monoxide (CO) levels to make sure they qualify for the trial. Participants will be asked to go to a nearby dentist who will look at their mouths. Participants will go back to the pharmacy and if they qualify, they will be given a supply of their assigned treatment. They will have an equal chance of receiving a treatment that has a drug in it or one that has no drug in it. They will be given a diary to keep track of how much of the treatment they use.

Subjects will go to the pharmacy four more times to hand in their diaries and blow into a machine that will measure their CO levels. At the last visit, subjects will have their mouths examined by a dentist again to have their mouth checked.

Subjects will receive four telephone calls during the study where they will be asked some questions.

After the 12 week treatment period, subjects will receive two to three more telephone calls, where they will be asked to answer some questions. Participants may be asked to come back to the pharmacy two more times to blow into the carbon monoxide machine again.

DETAILED DESCRIPTION:
This trial is a multi-center, randomized, double blind, placebo-controlled parallel group study to measure the efficacy and safety of a new nicotine replacement therapy for smoking cessation in a naturalistic environment. Subjects will be randomized in a 2:1 ratio (active to placebo). It is anticipated that data from about 450 in the active treatment group at Week 12 will be required for the safety analysis. In order to obtain that number of subjects, approximately 1500 subjects will need to be enrolled into the Use phase of the study, 1000 in the active arm and 500 in the placebo arm.

Based on the directions for use on the Drug Facts label, the study will include six weeks of full study drug treatment and then six weeks of progressive tapering drug treatment (Weeks 1-12). There will be a 14-week post-use follow up period.

This trial will be conducted in three sequential phases: Enrollment (baseline), Use and Post-use Follow-up. The Enrollment Phase will be conducted in approximately 20 pharmacies in nine diverse geographical areas in the continental United States. Subjects who qualify to participate in the study will be given three units of investigational product, a subject diary for tracking investigational product use and a medical problems worksheet to assist in the collection of AE information. Subjects will also be given a small hand counter and will be encouraged to use it to help keep track of the number of doses they use each day. Subjects will also be given a card with contact information for the pharmacy and study nurses. Where needed, the subject can also speak with the study physician.

During the Use Phase, the collection of data related to efficacy will be accomplished during four return visits to the pharmacy (at weeks 2, 4, 6 and 12). Self-reported abstinence will be verified by carbon monoxide (CO) measurements obtained at each pharmacy visit. Subjects will be given a subject use diary at each follow-up and re-supply visit and completed diaries will be collected each time the subject returns to the pharmacy. Subjects can return to the pharmacy for additional supplies at any time during their participation. Empty units will be returned during these visits.

Safety data will be collected during four telephone interviews, conducted by trained nurse interviewers, at weeks 2, 4, 6 and 12. If a subject reports an adverse event during a visit (return visit or resupply visit), this information will be immediately forwarded to the nurse interviewers for follow-up. Subjects may also initiate a call to the study nurses themselves to discuss health problems. All AE information collected will be reviewed by a physician as the adverse events are collected. A standardized visual mouth examination will be conducted by trained dentists at the enrollment visit and at the Week 12 return visit.

During the Post-use Follow-up period, self-reported efficacy and safety data will be collected during two telephone interviews initiated by trained nurse interviewers (at weeks 16 and 26). Subjects reporting abstinence since the last visit or abstinence for the prior seven days during these two interviews will be asked to return to the pharmacy to verify abstinence with an exhaled CO measurement. An additional telephone interview will be conducted between Week-12 and Week-16, by trained nurse interviewers, who will administer the End of Treatment questions to those subjects who have reported the following product use behavior that are inconsistent with the directions on the Drug Facts label: Use of more than 64 doses in a 24-hour period at least one time or use of more than 4 doses per hour at least one time based on the diary or their self report.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be males or females 18 years of age or older who currently smoke cigarettes and are willing to stop smoking

Exclusion Criteria:

* Subjects must not have a recent history of unstable angina, myocardial infarction or stroke
* They must not have a suspected malignant and/or erosive oral lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Qi, MD, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (19):
- United States (19):
  - Avalon Discount Drugs, Muscle Shoals, Alabama
  - Coast Compounding Pharmacy, Oceanside, California
  - Wynn's Pharmacy, Inc., Griffin, Georgia
  - Stark Pharmacy, Overland Park, Kansas
  - Goodrich Pharmacy, Anoka, Minnesota
  - Goodrich Pharmacy, Elk River, Minnesota
  - Goodrich Pharmacy, Saint Francis, Minnesota
  - Cub Pharmacy #1924, Saint Louis Park, Minnesota
  - Medicap Pharmacy, Clarksdale, Mississippi
  - Liddy's Health Mart, Holly Springs, Mississippi
  - Countryside Pharmacy, Savannah, Missouri
  - Phil's Pills, Albuquerque, New Mexico
  - Kerr Drug, Raleigh, North Carolina
  - Family Prescription Center, Bethlehem, Pennsylvania
  - T.B. Bond Pharmacy, Hillsboro, Texas
  - Inwood Pharmacy, Houston, Texas
  - Louis Morgan Drug #1, Longview, Texas
  - Brick Street Pharmacy, Tyler, Texas
  - Montpelier Pharmacy, Inc., Montpelier, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Nicotine
Started | 244 | 13
Completed | 0 | 0
Not Completed | 244 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 19 | 1
Not completed — Withdrawal by Subject | 12 | 0
Not completed — Difficulty Contacting Subject | 2 | 0
Not completed — Study Terminated by Sponsor | 209 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nicotine | Total
Number analyzed (Participants) | 244 | 13 | 257
Age Continuous [Mean (Standard Deviation); unit: years] | 47.1 (14.0) | 49.9 (11.4) | 47.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 8 | 139
  Male | 113 | 5 | 118
Region of Enrollment [Number; unit: participants]
  United States | 244 | 13 | 257

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Continuous Smoking Abstinence
Description: Number of participants with carbon monoxide (CO)-verified self-report of continuous abstinence from smoking from Week 2 through Week 6.
Time Frame: through Week 6
Population: The study was terminated prematurely due to a technical issue (randomization error) and no data are available.
Measure: Number; unit: Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Continuous Smoking Abstinence
Description: Number of participants with carbon monoxide (CO)-verified self report of continuous abstinence from smoking from Week 2 to Weeks 4, 6, 12, 16, and 26.
Time Frame: through Week 26
Population: The study was terminated prematurely due to a technical issue (randomization error) and no data are available.
Measure: Number; unit: Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With 7-day Point Prevalence Abstinence
Description: Number of participants with carbon monoxide (CO)-verified self-reported 7-day point prevalence abstinence from smoking at Weeks 2, 4, 6, 12, 16, and 26.
Time Frame: through Week 26
Population: The study was terminated prematurely due to a technical issue (randomization error).
Measure: Number; unit: Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Number of Daily Doses
Description: Mean number of daily doses by study week.
Time Frame: Week 1
Population: Analysis was limited to data collected from participants at Week 1.
Measure: Mean (Standard Deviation); unit: Daily Doses
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 142 | 6
Daily Doses | 16.7 (11.7) | 14.9 (7.3)

5. Secondary Outcome: Mean Number of Daily Doses
Description: Mean number of daily doses by study week.
Time Frame: Week 2
Population: Analysis was limited to data collected from participants at Week 2.
Measure: Mean (Standard Deviation); unit: Daily Doses
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 124 | 7
Daily Doses | 15.8 (11.4) | 18.0 (14.2)

6. Secondary Outcome: Mean Number of Daily Doses
Description: Mean number of daily doses by study week.
Time Frame: Week 3
Population: Analysis was limited to data collected from participants at Week 3.
Measure: Mean (Standard Deviation); unit: Daily Doses
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 76 | 5
Daily Doses | 13.1 (9.4) | 15.8 (9.2)

7. Secondary Outcome: Mean Number of Daily Doses
Description: Mean number of daily doses by study week.
Time Frame: Week 4
Population: Analysis was limited to data collected from participants at Week 4.
Measure: Mean (Standard Deviation); unit: Daily Doses
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 44 | 3
Daily Doses | 12.2 (10.8) | 10.5 (5.7)

8. Secondary Outcome: Mean Number of Daily Doses
Description: Mean number of daily doses by study week.
Time Frame: Week 5
Population: Analysis was limited to data collected from participants at Week 5.
Measure: Mean (Standard Deviation); unit: Daily Doses
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 21 | 1
Daily Doses | 10.9 (11.3) | 4.0 (0.0)

9. Secondary Outcome: Mean Number of Daily Doses
Description: Mean number of daily doses by study week.
Time Frame: Week 6
Population: Analysis was limited to data collected from participants at Week 6. Analysis of data for the remainder of the study weeks was not possible because the trial terminated prematurely due to a technical issue (randomization error).
Measure: Mean (Standard Deviation); unit: Daily Doses
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 5 | 0
Daily Doses | 13.3 (12.8) |

10. Secondary Outcome: Percentage of Participants With High Dosage
Description: Percentage of participants who used more than 64 doses in any one-day period.
Time Frame: within 12 Weeks
Population: Analysis was limited to data collected from participants who had used study medication at least one day.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 149 | 8
Percentage of Participants | 2.0 | 0

11. Secondary Outcome: Percentage of Participants With High Usage
Description: Percentage of participants who used more than four doses in any one-hour period.
Time Frame: within 12 Weeks
Population: Analysis was limited to data collected from participants who had used study medication at least one day.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 149 | 8
Percentage of Participants | 28.2 | 25

12. Secondary Outcome: Highest Rating of Desire/Urge to Smoke on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced the Desire/Urge to Smoke on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and who completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 2.2 | 0
  Somewhat | 30.4 | 100
  Moderately so | 33.7 | 0
  Very much so | 22.8 | 0
  Extremely so | 10.9 | 0

13. Secondary Outcome: Highest Rating of Irritability/Frustration/Anger on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced Irritability/Frustration/Anger on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and who completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 30.4 | 50.0
  Somewhat | 27.2 | 50.0
  Moderately so | 23.9 | 0
  Very much so | 15.2 | 0
  Extremely so | 3.3 | 0

14. Secondary Outcome: Highest Rating of Restlessness on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced Restlessness on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and who completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 43.5 | 0
  Somewhat | 25.0 | 100
  Moderately so | 12.0 | 0
  Very much so | 13.0 | 0
  Extremely so | 6.5 | 0

15. Secondary Outcome: Highest Rating of Difficulty Concentrating on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced Difficulty Concentrating on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 53.3 | 50.0
  Somewhat | 18.5 | 50.0
  Moderately so | 15.2 | 0
  Very much so | 9.8 | 0
  Extremely so | 3.3 | 0

16. Secondary Outcome: Highest Rating of Anxiety on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced Anxiety on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and who completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 44.6 | 50.0
  Somewhat | 23.9 | 0
  Moderately so | 15.2 | 0
  Very much so | 13.0 | 50.0
  Extremely so | 3.3 | 0

17. Secondary Outcome: Highest Rating of Dysphoric or Depressed Mood on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced Dysphoric or Depressed Mood on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and who completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 66.3 | 0
  Somewhat | 19.6 | 100
  Moderately so | 9.8 | 0
  Very much so | 3.3 | 0
  Extremely so | 1.1 | 0

18. Secondary Outcome: Highest Rating of Insomnia on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced Insomnia on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and who completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 56.5 | 50.0
  Somewhat | 22.8 | 0
  Moderately so | 10.9 | 50.0
  Very much so | 3.3 | 0
  Extremely so | 6.5 | 0

19. Secondary Outcome: Highest Rating of Increased Appetite on a Categorical Scale
Description: Participants are asked if during the last 24 hours they experienced Increased Appetite on a 5-grade categorical scale from Not at all to Extremely so.
Time Frame: within 12 Weeks
Population: Analysis was limited to participants who used study medication at least once and who completed the questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 92 | 2
Percentage of Participants
  Not at all | 54.3 | 0
  Somewhat | 13.0 | 100
  Moderately so | 15.2 | 0
  Very much so | 15.2 | 0
  Extremely so | 2.2 | 0

20. Secondary Outcome: Participant Score for General Perception of the Product
Description: Participants are asked to rate their general perception of the investigational product on a scale of 1-10, where 1=very poor and 10=excellent.
Time Frame: through Week 12
Population: The study was terminated prematurely due to a technical issue (randomization error) and no data are available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Participant Score for Product Effectiveness in Dealing With Cravings
Description: Participants are asked to rate the product in its effectiveness for dealing with cravings, on a scale of 1-5, where 1=not at all effective, and 5=extremely effective.
Time Frame: through 12 Weeks
Population: The study was terminated prematurely due to a technical issue (randomization error) and no data are available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Participant Score for Speed of Action
Description: Participants are asked to rate the product for speed of action, on a scale of 1-9, where 1=extremely slow and 9=extremely fast.
Time Frame: through 12 Weeks
Population: The study was terminated prematurely due to a technical issue (randomization error) and no data are available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Participant Score for Change in Perception
Description: Participants are asked to rate how their opinion has changed since the first time they used it, on a score of 1-5, where 1=I like it much less now and 5=I like it much more now.
Time Frame: through 12 Weeks
Population: The study was terminated prematurely due to a technical issue (randomization error) and no data are available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Participant Score for Product Convenience
Description: Participants are asked to rate how convenient the product is to use, on a scale of 1-5, where 1=not at all convenient and 5=extremely convenient.
Time Frame: through 12 Weeks
Population: The study was terminated prematurely due to a technical issue (randomization error) and no data are available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nicotine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during study and during telephone interview after study termination. Serious adverse events and adverse events categorized as probably or very likely related to study product were followed until they resolved or stabilized.
Description: Two subjects who did not receive study medication were excluded from the safety analysis set as defined in the Statistical Analysis Plan.
Arm/Group | Placebo | Nicotine
Serious Adverse Events (participants affected / at risk) | 4/242 | 1/13
Other Adverse Events (participants affected / at risk) | 33/242 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=242) | Nicotine (N=13)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Death (General disorders) | 1 | 0
Device Malfunction (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=242) | Nicotine (N=13)
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 1 | 1
Oral Pain (Gastrointestinal disorders) | 4 | 1
Sensitivity of Teeth (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 20 | 0
Migraine (Nervous system disorders) | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 5

LIMITATIONS AND CAVEATS:
Summary tabulations are not available for the primary and some secondary outcome measures because the study was terminated early due to a technical issue (randomization error).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators agreed not to discuss or publish the details/results of this study.